CLINICAL TRIAL: NCT06515977
Title: Impact of Texture and Color Enhancement Imaging on Detection and Miss Rate of Premalignant Lesions: A Multicentre, Randomized, Tandem Trial
Brief Title: Texture and Colour Enhancement Imaging in Improving Detection and Miss Rate of Premalignant Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); The Second Hospital of Hebei Medical University (Other); The Second Affiliated Hospital of Guangzhou University of Chinese Medicine (Unknown); Huadong Hospital (Other); Shanghai 6th People's Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); The General Hospital of Eastern Theater Command (Other); Jiangsu Provincial People's Hospital (Other); First People's Hospital of Hangzhou (Other); Wenzhou Central Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Shanxi Coal Center Hospital (Unknown); Dalian Municipal Central Hospital (Other); Seventh Medical Center of PLA Army General Hospital (Other); Henan Provincial People's Hospital (Other); Zunyi Medical College (Other); Shandong Second People's Hospital (Unknown); The Third People's Hospital of Chengdu (Other); Lanzhou University Second Hospital (Other); The Third People's Hospital of Jingdezhen (Unknown); Fudan University Attached Tumor Hospital (Unknown); Qingyuan People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: TADR-2024
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Adenoma; Sessile Serrated Adenoma
Keywords: texture and color enhancement imaging; colonoscopy; adenoma detection rate; sessile serrated lesion detection rate; adenoma miss rate; sessile serrated lesion miss rate
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TXI (Group A) (Experimental): Arm undergoing colonoscopy with TXI
  Interventions: Procedure: TXI (Group A)
- TXI followed by WLI (Group B) (Experimental): Arm undergoing initial inspection under TXI first, followed by second inspection with WLI
  Interventions: Procedure: TXI followed by WLI (Group B)
- WLI (Group C) (Active Comparator): Arm undergoing normal colonoscopy with WLI
  Interventions: Procedure: WLI (Group C)
- WLI followed by TXI (Group D) (Active Comparator): Arm undergoing initial inspection under WLI first, followed by second inspection with TXI
  Interventions: Procedure: WLI followed by TXI (Group D)

INTERVENTIONS:
Procedure: TXI (Group A) — Patients in Group A will undergo colonoscopy with TXI.
  Arms: TXI (Group A)
Procedure: TXI followed by WLI (Group B) — Patients in group B will first undergo colonoscopy with TXI and every polyp found should be removed. Then switch to WLI for a second withdrawal to detect lesions that were not observed the first time.
  Arms: TXI followed by WLI (Group B)
Procedure: WLI (Group C) — Patients in Group C will undergo colonoscopy with WLI.
  Arms: WLI (Group C)
Procedure: WLI followed by TXI (Group D) — Patients in group D will first undergo colonoscopy with WLI and every polyp found should be removed. Then switch to TXI for a second withdrawal to detect lesions that were not observed the first time.
  Arms: WLI followed by TXI (Group D)

SUMMARY:
Texture and Color Enhancement Imaging (TXI) is a newly developed image-enhancing endoscopy technology that has show potential in improving detection of colorectal lesions. This multicenter, randomized, tandem trial is aimed at evaluating whether TXI is superior to WLI endoscopy in terms of diagnosis of premalignant lesions.

ELIGIBILITY:
Inclusion Criteria:

patients aged 45-85 years and scheduled for screening colonoscopy who provided written informed consent

Exclusion Criteria:

Surveillance, diagnostic or therapeutic colonoscopy

Patients with an already known or suspected colorectal tumour

Patients with alarming symptoms and signs, including haematochezia, melena, weight loss or anaemia without specific causes, an abdominal mass and positive digital rectal examination

Pregnant or lactating women

Patients with gastrointestinal tract obstruction

Patients with inflammatory bowel diseases, hereditary CRC syndromes or serrated polyposis syndrome

Patients with abnormal blood coagulation or taking antiplatelets or anticoagulants within 7 days before colonoscopy

Patients with failed cecal intubation

Patients with poor bowel preparation quality that necessitated a second bowel preparation

Patients with a history of colonic resection

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2964 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
adenoma detection rate | 1 years
  the number of patients with one or more adenomas detected and removed divided by the total number of patient
sessile serrated lesion detection rate | 1 years
  the number of patients with one or more sessile serrated lesions detected and removed divided by the total number of patients

SECONDARY OUTCOMES:
adenoma miss rate | 1 years
  the number of adenomas detected during the second examination divided by the total number of adenomas detected during the first and second colonoscopy
sessile serrated lesion miss rate | 1 years
  the number of sessile serrated lesions detected during the second examination divided by the total number of sessile serrated lesions detected during the first and second colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital

REFERENCES:
- [Background] Wei J, Zhao S, Bai Y. Impact of Texture and Color Enhancement Imaging on Adenoma and Sessile Serrated Lesion Detection: Much More to Explore. Gastroenterology. 2024 Jul;167(2):413-414. doi: 10.1053/j.gastro.2024.01.014. Epub 2024 Jan 13. No abstract available. PMID 38224857
- [Background] Antonelli G, Bevivino G, Pecere S, Ebigbo A, Cereatti F, Akizue N, Di Fonzo M, Coppola M, Barbaro F, Walter BM, Sharma P, Caruso A, Okimoto K, Antenucci C, Matsumura T, Zerboni G, Grossi C, Meinikheim M, Papparella LG, Correale L, Costamagna G, Repici A, Spada C, Messmann H, Hassan C, Iacopini F. Texture and color enhancement imaging versus high definition white-light endoscopy for detection of colorectal neoplasia: a randomized trial. Endoscopy. 2023 Dec;55(12):1072-1080. doi: 10.1055/a-2129-7254. Epub 2023 Jul 14. PMID 37451283
- [Background] Young E, Rajagopalan A, Tee D, Sathananthan D, Hoile S, Singh R. Texture and Color Enhancement Imaging Improves Colonic Adenoma Detection: A Multicenter Randomized Controlled Trial. Gastroenterology. 2024 Feb;166(2):338-340.e3. doi: 10.1053/j.gastro.2023.10.008. Epub 2023 Oct 14. PMID 37839498